CLINICAL TRIAL: NCT07217626
Title: Pre-Incision Peripheral Nerve Blocks Versus No Peripheral Nerve Blocks for Lower Extremity Fracture Surgery in Older Adults: A Pilot Feasibility Study
Brief Title: Pre-Incision Peripheral Nerve Blocks for Lower Extremity Fracture Surgery in Older Adults
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Arissa Torrie, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HP-00115610
Record Dates: First submitted 2025-10-03; First posted 2025-10-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Lower Extremity Fracture; Surgical Fracture Repair; Orthopaedic Trauma; Orthogeriatric Fractures
Keywords: Regional Anesthesia; Clinical Outcomes; Orthopaedic trauma; Perioperative Outcomes; Pilot Study; Lower Extremity Fractures; Orthogeriatric Fractures; Peripheral Nerve Blocks

STUDY DESIGN:
Intervention Model Description: Pilot Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-incision Peripheral Nerve Blocks (Active Comparator): Long-acting local anesthesia for pre-incision peripheral nerve blocks that cover the fracture and surgical pain during definitive surgical fixation of lower extremity fractures.
  Interventions: Drug: Local anesthesia injections
- No peripheral nerve block (No Intervention): No peripheral nerve block for definitive surgical fixation of lower extremity fractures. Participants can receive standard anesthesia options for their surgical intervention including neuraxial or general anesthesia, surgical site infiltration, and multimodal analgesia.

INTERVENTIONS:
Drug: Local anesthesia injections — The peripheral nerve block should be performed within 2 hours before incision, either in the pre-operative holding area when called to the operating room or after positioning but prior to skin antisepsis in the operating room. The goal is to achieve an established neural blockade before surgical incision without delaying the surgical start time. All blocks must be performed using ultrasound guidance. Consistent with clinical practice, anesthesiologists will determine the appropriate balance between motor and sensory blockade based on patient factors, surgical approach, and clinical judgment.
  Other Names: peripheral nerve block
  Arms: Pre-incision Peripheral Nerve Blocks

SUMMARY:
Fractures of the lower leg are especially difficult for older adults. They are more likely to have serious complications, require longer healing times, and have a higher risk of death This occurs because their bodies cannot tolerate stress as well as younger individuals. The injury itself places significant strain on the body, and surgery adds additional stress.

Anesthesiologists use nerve blocks to help manage pain during and after these injuries. A nerve block is an injection that numbs the fracture and surgery area by blocking pain signals. These injections help patients need fewer opioid medications. However, new research shows these nerve blocks may provide benefits beyond pain management. Studies looking at older adults with hip fractures who received nerve blocks showed better overall outcomes: fewer deaths, fewer serious complications, and shorter hospital stays.

However, it is not currently known if nerve blocks work this well for other broken bones in the leg, like in the thigh or shin. Additional research is need to know if nerve blocks can help patients with all types of leg fractures recover faster and experience fewer problems.

Before the investigators start a large clinical trial, a small pilot study needs to be completed to determine if a larger clinical trial is feasible. This pilot study will evaluate the ability to recruit enough patients, ensure patients can receive the assigned treatment, collect data effectively, follow the study protocol, and track participants over time. The results will indicate whether the investigators are prepared to proceed with a full-scale trial and help refine the approach.

DETAILED DESCRIPTION:
The potential for peripheral nerve blocks to improve clinical outcomes beyond analgesia is based on their ability to interrupt the physiologic stress response to surgical trauma near its origin. Tissue injury triggers nociceptive signals that travel through peripheral nerves to initiate a cascade of neuroendocrine and inflammatory responses, including the release of catecholamines, activation of the hypothalamic-pituitary-adrenal axis, and systemic inflammation. While younger patients can tolerate this stress response, older adults with limited physiologic reserve may experience organ dysfunction when these compensatory mechanisms become overwhelmed. By blocking afferent neural transmission before it reaches the central nervous system, peripheral nerve blocks may attenuate this cascade, potentially reducing sympathetic surge, myocardial oxygen demand, and the release of inflammatory mediators. Additionally, effective peripheral nerve blocks can reduce opioid requirements, avoiding adverse effects including respiratory depression, delirium, and impaired mobilization that particularly affect older adults. These mechanistic advantages may be especially important in older adults with lower extremity fractures, who face both the initial trauma and the additional physiologic burden of surgical repair.

While peripheral nerve blocks are well-established components of multimodal analgesia, emerging evidence suggests their benefits may extend beyond short-term analgesic effects. Recent studies of older adults with hip fractures have found peripheral nerve blocks are associated with additional benefits including reduced mortality, fewer serious adverse events, and increased days alive out of hospital. However, evidence for fractures distal to the hip remains limited. Although current Orthopaedic Trauma Association guidelines recommend peripheral nerve blocks as part of multimodal pain management for hip fractures, time pressures, and uncertainty about benefits beyond short-term analgesia have resulted in variable adoption among anesthesiologists and orthopaedic surgeons. Evidence supporting broader use of peripheral nerve blocks for improving clinical outcomes in lower extremity fractures is still needed.

To address this knowledge gap, a large multicenter randomized controlled trial is needed. However, prior to initiating such a trial, a pilot feasibility study will be conducted comparing pre-incision peripheral nerve blocks to no peripheral nerve blocks. The primary objective is to assess feasibility in terms of patient recruitment, adherence to treatment allocation, data collection methods, protocol compliance, and participant follow-up. This pilot phase will allow for refinement of the primary outcome measure, optimization of data collection procedures, establishment of recruitment rates, and identification of potential barriers to implementation before committing resources to a large-scale definitive trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years
2. Isolated fractures
3. Radiographically confirmed lower extremity fracture requiring surgical fixation including:

   1. Femoral shaft
   2. Distal femur
   3. Patella
   4. Proximal tibia
   5. Tibial shaft
   6. Distal Tibia
   7. Pilon fractures
   8. Ankle (malleolar fractures)
   9. Calcaneus
   10. Talus
   11. Hindfoot/midfoot
4. Acute fracture receiving definitive fixation during injury hospitalization

4) Ability to provide informed consent (patient or legally authorized representative (LAR))

Exclusion Criteria:

1. Contraindication to peripheral nerve block

   1. Infection at planned needle insertion site
   2. Patient refusal
   3. Surgeon or anesthesiologist refusal secondary to the patient's medical status
2. Active peripheral nerve blockade from initial injury analgesic management is defined as:

   a. Risk of local anesthetic systemic toxicity
3. Neurologic or vascular injuries in the affected limb
4. Polytrauma with traumatic brain injury
5. Thoracic injury and/or abdominal injury requiring surgical intervention
6. Current enrollment in a conflicting clinical trial
7. Acute or Subacute residence prior to injury
8. Incarcerated at the time of enrollment
9. Prior enrollment in this trial
10. Unable to obtain informed consent due to language barrier
11. Unable to obtain informed consent because a legally authorized representative was unavailable.
12. Anticipated problems with follow-up compliance

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Participant Enrollment | 12 months
  Participant enrollment will be assessed by monitoring screening and enrollment metrics, including:
  * Initiation of screening and recruitment at the clinical site
  * Ability of the clinical site to screen consecutive patients 50 years of age and older with lower extremity fractures
  * Proportion of patients who are screened for eligibility to participate in the trial
  * Proportion of patients who meet the eligibility criteria
  * Review of reasons for exclusion
  * Proportion of patients who provide informed consent
  * Length of time required to enroll up to 50 patients
Feasibility of Treatment Allocation | 12 months
  Feasibility of the treatment allocation will be assessed using the following metrics:
  * Proportion of adherence to pre-incision peripheral nerve block allocation
  * Proportion of adherence to no peripheral nerve block allocation
  * Proportion of stage 2 consent acceptance rate among participants randomized to peripheral nerve blocks
Refine Data Collection Methods | 12 months
  To refine the data collection methods, the following metrics will be reviewed:
  * Proportion of participants with missing data
  * Proportion of missing data to identify data fields that are not feasible to collect
  * Proportion of data errors to identify ways to improve the flow of the case report forms (CRFs) and data collection
Assess Protocol Compliance | Day 30 + 5 post-randomization
  The following metrics will be used to assess compliance with the protocol:
  * Proportion of randomization errors
  * Proportion of participants who complete the 30-day follow-up phone call
  * Proportion of participants who withdraw from the trial (withdrawal of consent)
  * Proportion of participants who cannot be located (loss to follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Arissa Torrie, MD, MHS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: The results of this pilot feasibility study protocol will be published on an open-access peer-reviewed journal.
Access Criteria: The results of this pilot feasibility study protocol will be published on an open-access peer-reviewed journal.